CLINICAL TRIAL: NCT02083549
Title: Evaluating the Efficacy of the University of Rochester Medical Center's Massive Transfusion Protocol in Trauma Level 1 Patients Utilizing Thromboelastography
Brief Title: Evaluating URMC's Massive Transfusion Protocol
Acronym: MTP-TEG
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Majed Refaai, Associate Professor, University of Rochester
Other Study IDs: UR- MTP-TEG
Record Dates: First submitted 2014-03-05; First posted 2014-03-11 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Blood Coagulation Disorders; Trauma; Acute Coagulopathy
Keywords: Massive Transfusion Protocol
MeSH Terms: conditions — Blood Coagulation Disorders; Wounds and Injuries | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Trauma 1 massively transfused: Trauma 1 massively transfused patients are identified as a Trauma level one patient by triage through guidelines from the Kessler Regional Trauma Center Trauma Triage Guidelines.
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: Blood collection — After transfusion of each shipment of blood products outlined in the current Massive Transfusion Protocol one 2.7mL citrated blood sample will be collected from the subject through the 5th shipment of blood products. A final sample will be collected 24 hours following the discontinuation of the massive transfusion protocol.

SUMMARY:
The purpose of the study is to evaluate the efficacy of the University of Rochester Medical Center's current Massive Transfusion Protocol.

Upon arrival of trauma level one designated patients the treating team evaluates the patient's injuries. If the patient is initiated under the facilities Massive Transfusion Protocol and meets other inclusion and exclusion criteria the patient will be enrolled in the study. Study procedures include collection of a blood sample following the transfusion of each shipment, through shipment 5, of blood products outlined in the current Massive Transfusion Protocol.

Each blood sample will be run on a Thromboelastograph to evaluate the patient's hematostatic state through resuscitation. One final blood sample will be collected 24 hours following the discontinuation of the Massive Transfusion Protocol and also ran on the thromboelastograph.

Due to the critical need for medical intervention, consent procedure will be waived at time of enrollment. An authorized representative for the patient will be identified and approached to obtain consent for use of data collected.

ELIGIBILITY:
Inclusion Criteria:

* Trauma level 1 patient initiated under Massive Transfusion Protocol
* Age greater than or equal to 18 years old

Exclusion Criteria:

* Females who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes level 1 trauma patients brought to the trauma bay for resusitation and are initiated under the Massive Transfusion Protocol.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2014-12-16 (Actual); Study Completion 2014-12-16 (Actual)

PRIMARY OUTCOMES:
Efficacy of Blood product ratio | 24 hours
  Through thromboelastography testing the coagulopathy of trauma 1 patients receiving massive amounts of blood products in a ratio previously established by the institutions Standard of Procedure will be evaluated to determine the efficacy of the current blood product ratio.

SECONDARY OUTCOMES:
Haemostasis clot kinetics | 24 hours
  Kinetics of clot formation analyzed by thromboelastograph over the course of the first 24 hours of resuscitation.

OTHER OUTCOMES:
Standard clinical data | 24 hours
  Patient and trauma specific information will be extracted from the patients' record. Including but not limited to age, gender, type of injury and severity score, assessment of blood consumption score, blood type, number and volume of blood transfusions consumed during present trauma, current and past medical history and medications.

CONTACTS AND LOCATIONS:
Overall Officials: Majed Refaai, MD, Principal Investigator — University of Rochester
Locations (1):
- Strong Hospital at University of Rochester Medical Center, Rochester, New York, United States